CLINICAL TRIAL: NCT01658657
Title: A Pilot Study of Plasma Renin Activity Guided vs Generic Combination Therapy for Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Cornell University (Other); Wake Forest University Health Sciences (Other)
Responsible Party: Principal Investigator, Anthony J Viera, MD, MPH, Distinguished Associate Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12-1133
Record Dates: First submitted 2012-07-31; First posted 2012-08-07 (Estimated); Results first posted 2015-06-22 (Estimated); Last update posted 2015-08-27 (Estimated); Status verified 2015-08

CONDITIONS: Hypertension; Plasma Renin Activity
MeSH Terms: conditions — Hypertension | interventions — Hydrochlorothiazide; Lisinopril; Amlodipine; Metoprolol; hydrochlorothiazide, lisinopril drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- PRA-guided therapy (Experimental): Participants randomized to the PRA-guided therapy treatment arm will be prescribed anti-hypertensive medications based on renin activity level as defined at baseline.
  Interventions: Drug: Hydrochlorothiazide; Drug: Lisinopril; Drug: Amlodipine; Drug: metoprolol
- Fixed-dose combination treatment-guided therapy (Active Comparator): Participants randomized to the fixed-dose combination treatment-guided arm will be prescribed standard anti-hypertensive medications without regard to renin activity level.
  Interventions: Drug: Amlodipine; Drug: metoprolol; Drug: lisinopril/hydrochlorothiazide

INTERVENTIONS:
Drug: Hydrochlorothiazide
  Arms: PRA-guided therapy
Drug: Lisinopril
  Arms: PRA-guided therapy
Drug: Amlodipine
Drug: metoprolol
Drug: lisinopril/hydrochlorothiazide — This is a combination pill
  Arms: Fixed-dose combination treatment-guided therapy

SUMMARY:
The purpose of this study is to investigate the effect of plasma renin activity-guided therapy for determining hypertension treatment. Plasma renin is an enzyme in your blood that can be measured to determine your hypertension subtype. Once the subtype is known, doctors can prescribe specific medications to target your specific hypertension subtype. This study will investigate whether targeting the specific hypertension subtype helps to achieve blood pressure control sooner and with fewer medications compared to a standard fixed dose combination therapy.

ELIGIBILITY:
Inclusion Criteria:

* Systolic BP average during at least one recent (within 1 month) clinic or emergency room visit ≥ 150 mmHg, or diastolic BP average during at least one recent (within 1 month) clinic or emergency room visit ≥ 95 mmHg
* Not currently taking BP-lowering medication
* Clinician recommends pharmacologic treatment
* Willing to make necessary study visits
* Able to be contacted by phone
* Has a primary care clinician
* At least 18 years old

Exclusion Criteria:

* Known secondary cause of hypertension
* Pregnancy
* Known diabetes, coronary artery disease or renal disease
* Known sulfonamide allergy or history of gout
* Participant's clinician recommends he/she not enroll
* Hyponatremia, hypokalemia, hypernatremia, or hyperglycemia at baseline visit
* Baseline visit systolic visit BP average < 140 mmHg and diastolic BP average < 90 mm Hg
* Resting heart rate < 55 beats per minute

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2012-10; Primary Completion 2014-07 (Actual); Study Completion 2014-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Viera, MD, MPH, Principal Investigator — Distinguished Associate Professor, Family Medicine
Locations (1):
- UNC Chapel Hill, Chapel Hill, North Carolina, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- PRA-guided Therapy: Participants randomized to the PRA-guided therapy treatment arm will be prescribed anti-hypertensive medications based on renin activity level as defined at baseline.
  Hydrochlorothiazide
  Lisinopril
  Amlodipine
  metoprolol
- Fixed-dose Combination Treatment-guided Therapy: Participants randomized to the fixed-dose combination treatment-guided arm will be prescribed standard anti-hypertensive medications without regard to renin activity level.
  Amlodipine
  metoprolol
  lisinopril/hydrochlorothiazide
Period: Overall Study
Arm/Group | PRA-guided Therapy | Fixed-dose Combination Treatment-guided Therapy
Started | 7 | 10
Completed | 4 | 7
Not Completed | 3 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PRA-guided Therapy | Fixed-dose Combination Treatment-guided Therapy | Total
Number analyzed (Participants) | 7 | 10 | 17
Age, Continuous [Mean (Full Range); unit: years] | 47.6 [35 to 59] | 46.7 [27 to 67] | 47 [27 to 67]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 5 | 5 | 10
Region of Enrollment [Number; unit: participants]
  United States | 7 | 10 | 17

OUTCOME MEASURES:

1. Primary Outcome: Blood Pressure Control, as Defined as Office BP Measurement of <140 mmHg Systolic and <90 mmHg Diastolic
Description: At each study visit (approximately every 30 days), participants' BP will be checked. If BP is controlled (<140mmHG systolic and <90mmHG diastolic), then current medication will continue. If BP is uncontrolled, medication will be revised every 30 days (up to 120) until BP control is achieved.
Time Frame: 4 months
Population: 6 participants withdrawn before study completion
Measure: Number; unit: participants
Arm/Group | PRA-guided Therapy | Fixed-dose Combination Treatment-guided Therapy
Number analyzed (Participants) | 4 | 7
participants | 3 | 1

ADVERSE EVENTS:
Arm/Group | PRA-guided Therapy | Fixed-dose Combination Treatment-guided Therapy
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/10
Other Adverse Events (participants affected / at risk) | 3/7 | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PRA-guided Therapy (N=7) | Fixed-dose Combination Treatment-guided Therapy (N=10)
Electrolyte disturbance (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Lightheadedness (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No